CLINICAL TRIAL: NCT03858517
Title: A Post-Market Clinical Evaluation of the ReUnion TSA System
Status: Terminated | Type: Observational
Why Stopped: Sponsor Terminated
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: ReUnion TSA Study
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ReUnion TSA System: Subject with one or more of the following diagnoses will be treated with the ReUnion TSA System:
  * Aseptic necrosis of the humeral head
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis, rheumatoid arthritis or post-traumatic arthritis
  * Failed previous total shoulder replacement, resurfacing or other procedure
  Interventions: Device: ReUnion TSA System

INTERVENTIONS:
Device: ReUnion TSA System — The ReUnion TSA System is designed as an anatomical total shoulder or hemi-shoulder endoprosthesis to address advanced arthritic disorders affecting the shoulder joint in subjects having intact or repairable rotator cuff function. The ReUnion TSA System consists of a completely modular shoulder platform including a Humeral Stem, Humeral Head and Glenoid. The intended purposes of the ReUnion TSA System are to achieve pain relief, improvement of range of motion and restoration or improvement of the shoulder function while ensuring long-term replacement of the shoulder joint with sufficient stability of all endoprosthesis components.

SUMMARY:
This investigation is a prospective, multicenter clinical investigation. It is anticipated that a total of one hundred (100) subjects will be enrolled at approximately 4-7 sites. The clinical investigation has been designed to follow the surgeon's standard of care for joint arthroplasty subjects, which entails clinical evaluation on a regular ongoing basis, or as needed should the subject become symptomatic in the treated joint.

DETAILED DESCRIPTION:
The objective of this clinical investigation is to demonstrate the safety and efficacy/performance of the ReUnion TSA System. Efficacy/performance of the procedure will be measured the American Shoulder and Elbow Surgeons (ASES) Shoulder Score. Safety of the ReUnion TSA System will be demonstrated through reporting of device-related intra-operative and post-operative Adverse Events (AEs). Enrolled subjects will be assessed at Pre-Operative, Operative/Discharge, and at 6 Weeks, 6 Months, 12 Months, 24 Months and annually thereafter up to 10 years following the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to sign the informed consent.
* Subject is willing and able to comply with postoperative scheduled clinical and radiographic evaluations.
* Subject is male or non-pregnant female and 18 years or older at the time of surgery.
* Subject has one or more of the following:

  * Aseptic necrosis of the humeral head
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis, rheumatoid arthritis or post-traumatic arthritis
  * Failed previous total shoulder replacement, resurfacing or other procedure

Exclusion Criteria:

* Subject has an active or suspected latent infection in or about the shoulder joint.
* Subject has mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure or complications in postoperative care.
* Subject has bone stock compromised by disease, infection or prior implantation which cannot provide adequate support and/or fixation to the prosthesis.
* Subject has anticipated activities which would impose high stresses on the prosthesis and its fixation.
* Subject is obese such that he/she produces a load on the prosthesis which can lead to failure of fixation of the device or to failure of the device itself.
* Subject has absent, irreparable or non-functioning rotator cuff and other essential muscles.
* Subject has concomitant disease(s) which may significantly affect the clinical outcome.
* Subject has traumatic or pathologic fracture of the proximal humerus.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 subjects are to be enrolled in this clinical investigation. The clinical investigation has been designed to follow the surgeon's standard of care for joint arthroplasty subjects, which entails clinical evaluation on a regular ongoing basis, or as needed should the subject become symptomatic in the treated joint.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma
Locations (3):
- United States (3):
  - Great Plains Orthopedics, Peoria, Illinois
  - Tennessee Orthopaedic Alliance, Nashville, Michigan
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ReUnion TSA System: Subject with one or more of the following diagnoses will be treated with the ReUnion TSA System:
  * Aseptic necrosis of the humeral head
  * Painful, disabling joint disease of the shoulder resulting from degenerative arthritis, rheumatoid arthritis or post-traumatic arthritis
  * Failed previous total shoulder replacement, resurfacing or other procedure
  ReUnion TSA System: The ReUnion TSA System is designed as an anatomical total shoulder or hemi-shoulder endoprosthesis to address advanced arthritic disorders affecting the shoulder joint in subjects having intact or repairable rotator cuff function. The ReUnion TSA System consists of a completely modular shoulder platform including a Humeral Stem, Humeral Head and Glenoid. The intended purposes of the ReUnion TSA System are to achieve pain relief, improvement of range of motion and restoration or improvement of the shoulder function while ensuring long-term replacement of the shoulder joint with sufficient stability of all endoprosthesis components.
Period: Overall Study
Arm/Group | ReUnion TSA System
Started | 51
Completed | 0
Not Completed | 51
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — removed for being incarcerated | 1
Not completed — Sponsor Closure | 48

BASELINE CHARACTERISTICS:
Arm/Group | ReUnion TSA System
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.08 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Black or African | 2
  Ethnicity: Native Hawaiian or Other Pacific Islander | 1
  Ethnicity: Caucasian | 46
  Ethnicity: Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 32.29 (5.56)

OUTCOME MEASURES:

1. Primary Outcome: American Shoulder and Elbow Surgeons (ASES) Shoulder Score
Description: The primary endpoint of the clinical investigation is to demonstrate non-inferiority of the device to the selected literature controls, as measured by the ASES Shoulder Score at 24 Months post-operative. Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
Time Frame: 24 months
Population: The Total ASES Shoulder Score (1 & 2 year LOCF) was available for 24 subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ReUnion TSA System
Number analyzed (Participants) | 24
score on a scale | 78.75 (26.19)

2. Secondary Outcome: Safety Will be Measured by Capturing the Incidence Rate of Device-related Intra-operative and Post-operative Adverse Events Will be Measured.
Description: Secondary outcome measures to assess safety by capturing the incidence rate of device-related intra-operative adverse events.
Time Frame: 24 mths
Population: 5 out of 51 Subjects with reportable Adverse Events. Please see Adverse Events section for break-down.
Measure: Count of Participants; unit: Participants
Arm/Group | ReUnion TSA System
Number analyzed (Participants) | 51
Participants | 5

3. Secondary Outcome: Efficacy Will be Measured by Monitoring All Implant Survivorship in All Subjects Who Have the Total or Partial Prosthesis With Full or Partial Implant Survival.
Description: Secondary outcome measures to assess efficacy by monitoring all implant survivorship in all subjects enrolled who have the ReUnion RFX System.
Time Frame: From Baseline to last recorded follow-up (~27 Months)
Population: 2 out of 51 Subjects had this data available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ReUnion TSA System
Number analyzed (Participants) | 2
days | 750.24 (37.09)

ADVERSE EVENTS:
Time Frame: From Baseline until study was terminated early (~27 Months).
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | ReUnion TSA System
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 5/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ReUnion TSA System (N=51)
Implant breakage/wear, humeral or glenoidal (Product Issues) | 1
Nerve injury, mild (minor motor or sensory loss, or spontaneous recovery) (Nervous system disorders) | 1
Nerve injury, severe (significant motor or sensory loss or requiring surgical revision) (Nervous system disorders) | 1
Rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1
Stiffness (Musculoskeletal and connective tissue disorders) | 1

LIMITATIONS AND CAVEATS:
As the study was terminated early, outcomes and adverse events can only be reported up to the date of closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03858517/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT03858517/SAP_001.pdf